CLINICAL TRIAL: NCT03334474
Title: Shnaghai Shengkang Medical Center
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guoxiang Fu (Other)
Responsible Party: Sponsor-Investigator, Guoxiang Fu, Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Organization: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Other Study IDs: shengkang
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- young: 18-35 years old
- middle: 35-65 years old
- aged: 65-85 years old

INTERVENTIONS:
Other:  — no intervention

SUMMARY:
The process of population aging that is occurring in developed societies represents a major challenge for the health system. The aim of this study is to analyze factors that have an influence on early vascular aging (EVA), estimated by carotid-femoral pulse wave velocity (cf-PWV) and Cardio Ankle Vascular Index (CAVI), and to determine differences by gender in a Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 35 to 85 years who agree to participate in the study and do not meet any of the exclusion criteria.

Exclusion Criteria:

* • Subjects who are in terminal condition, who cannot travel to the health centers to undergo the corresponding examinations, and those who do not wish to sign the informed consent.

  * Subjects with a history of CVD (ischemic heart disease or stroke, peripheral arterial disease or heart failure), diagnosed renal failure in terminal stages (glomerular filtration rate below 30%), chronic inflammatory disease, or acute inflammatory process in the past three months.
  * Patients treated with estrogens, testosterone, or growth hormone.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population It will be the urban population attached to the Health Center of Shanghai. Using a random sampling stratified by age groups and gender, 300 subjects will be selected in each group (150 males and 150 females), aged 35 to 85 years.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Cardio-ankle vascular index | 2 years
  This parameter will be estimated using Vasera device VS-1500.

IPD SHARING:
Plan to Share IPD: No